CLINICAL TRIAL: NCT02896010
Title: Effectiveness of a Personalized Smartphone-assisted Coaching System to Improve Glucose Homeostasis in Adults With Prediabetes: Rationale and Study Protocol - Pilot Study
Brief Title: Personalized Smartphone-assisted Coaching System to Improve Glucose Homeostasis in Adults With Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Sweetch Health, Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00099812
Record Dates: First submitted 2016-08-01; First posted 2016-09-12 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Prediabetes; Hyperglycemia; Postprandial Hyperglycemia; Impaired Glucose Tolerance; Impaired Fasting Glucose
Keywords: Mobile Health
MeSH Terms: conditions — Prediabetic State; Hyperglycemia; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sweetch App + DBWS (Active Comparator): Participants receive usual care for prediabetes management. In addition, participants will be randomized to receive the Sweetch app plus weight monitoring via digital body weight scale (DBWS).
  Interventions: Other: Sweetch App + DBWS
- Sweetch App Alone (Active Comparator): Participants receive usual care for prediabetes management. In addition, participants will be randomized to receive the Sweetch app alone.
  Interventions: Other: Sweetch App Alone

INTERVENTIONS:
Other: Sweetch App + DBWS — Usual care for prediabetes management, Sweetch app, weight monitoring via digital body weight scale (DBWS).
  Arms: Sweetch App + DBWS
Other: Sweetch App Alone — Usual care for prediabetes management, Sweetch app alone.
  Arms: Sweetch App Alone

SUMMARY:
Sweetch is a personalized mobile-health platform coaching system (mobile phone app) designed to promote adherence to physical activity guidelines for people with prediabetes.

DETAILED DESCRIPTION:
The mobile phone app Sweetch seeks to increase leisure time physical activity rather than formal exercise through the use of a behavioral analytics engine that continuously process various aspects of the user's life habits, taking into account the user's demographics, behavioral change status, schedule, actual activity patterns, and more. The rationale behind this approach is that long-term adherence and patient engagement are more likely to be achieved when demands on manual user data entry are kept at a minimum. Compared to similar smartphone-assisted prevention apps, there are two novel features of the Sweetch app that may increase its efficacy. First, it uses a "just-in-time" adaptive intervention" approach that tailors recommendations to the user's day-to-day routine and his or her readiness for behavioral change. Second, and most importantly, it requires no direct involvement by the user, since all the necessary data is collected using built-in tracking pedometers, accelerometer and GPS (Global Positioning System) sensors on smartphones. In contrast, interventions that focus on dietary changes (i.e. calorie reduction, change in macronutrient content), require active user tracking at every meal, which is difficult to maintain in the long-term even with the use of sophisticated, electronic calorie counting tools. For these reasons, the Sweetch app may achieve greater long-term adherence, which is usually a limiting factor to efficacy of mobile health interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 -75 years with prediabetes (fasting BG 100-125 mg/dl, A1C 5.7% - 6.4%, or 2 hour BG of 140-199 mg/dl following 75-gram oral glucose tolerance test)
* Body mass index 24 - 40 kg/m2
* English speaker
* Smartphone user (Android or Apple 5s and above)

Exclusion Criteria:

* Currently doing more than 150 minutes/week of moderate/vigorous physical activity
* Presence of medical conditions that prevent adoption of moderate physical activity
* Use of any glucose-lowering or weight loss medications within the previous 3 months
* Current pregnancy (self-reported) or planning pregnancy during study period (self-reported)
* Presence of any condition that can result in spurious A1C readings (e.g. anemia [hemoglobin level below lower limit of normal] secondary to iron, vitamin B12, or folate deficiencies; hemoglobinopathies)
* Use of systemic glucocorticoids
* Use of antipsychotic medications (stable doses for at least three months of anti-depressants or anti-anxiety drugs will be allowed)
* Severe mental illness or learning disability
* Current participation in another clinical trial
* Liver enzymes >3 x upper limit of normal
* Poor literacy (REALM-R score of 6 or less)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
Yield of Recruitment | 3 months
  Proportion of recruited participants who enroll and complete the 3 month study

SECONDARY OUTCOMES:
Engagement | 3 months
  Proportion of enrolled participants who keep app installed and open in background of their smartphones during duration of the study.
Usability and Satisfaction | 3 months
  Usability and Satisfaction will be measured using an adapted Systems Usability Scale, a validated method of measuring usability with a wide array of technological products, including smartphones.
Adherence to physical activity goal | 3 months
  Proportion of enrolled participants meeting mean 150 minute per week physical activity target (evaluated at 4 week intervals and over course of entire 12 week study period)

CONTACTS AND LOCATIONS:
Overall Officials: Nestoras Mathioudakis, MD MHS, Principal Investigator — Johns Hopkins University; Adrian S Dobs, MD MHS, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Reading Health System, Reading, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Everett E, Kane B, Yoo A, Dobs A, Mathioudakis N. A Novel Approach for Fully Automated, Personalized Health Coaching for Adults with Prediabetes: Pilot Clinical Trial. J Med Internet Res. 2018 Feb 27;20(2):e72. doi: 10.2196/jmir.9723. PMID 29487046